CLINICAL TRIAL: NCT05510583
Title: Non Inferiority Study of Glycemic Monitoring Via MyDiabby Healthcare Vs Conventional Diary in Patients with Gestational Diabetes Mellitus
Brief Title: MyDiabby Healthcare Vs Diary in Gestational Diabetes Mellitus.
Acronym: TELESUR-GDM
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD2421
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-05

CONDITIONS: Gestational Diabetes
Keywords: diabetes mellitus; tele-medicine; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Pregnant women (≥18 years) with gestational diabetes who gave birth between 01/01/2013 and 30/06/2015. Patients received traditional paper-based blood glucose monitoring.
  Interventions: Other: Control group
- Group 2: Pregnant women (≥18 years) with gestational diabetes who gave birth between 01/01/2021 and 31/12/2021. Patients received remote monitoring with myDiabby Healthcare
  Interventions: Other: Treated group

INTERVENTIONS:
Other: Control group — Retrospective study on pregnant women (≥18 years) with gestational diabetes who gave birth between 01/01/2013 and 30/06/2015. Patients received traditional paper-based blood glucose monitoring.
  Groups: Group 1
Other: Treated group — Retrospective study on pregnant women (≥18 years) with gestational diabetes who gave birth between 01/01/2021 and 31/12/2021. Patients received remote monitoring with myDiabby Healthcare
  Groups: Group 2

SUMMARY:
The purpose of the study is to demonstrate the non-inferiority of the onset of maternal, foetal, and neonatal complications for patients who had Gestational diabetes mellitus (GDM) and who had been monitored by myDiabby Healthcare compared to patients who had a classic glycemic blood monitoring by diary

DETAILED DESCRIPTION:
TELESUR-GDM is a descriptive and comparative study which will be compared to ERD2 study. ERD2 (personal data) was a retrospective study leaded in Rene Dubos hospital. The primary objective was to evaluate de proportion of patients who had a blood screening for type 2 diabetes after having a gestational diabetes and who gave birth between 2013 and 2015 in Rene Dubos hospital. The primary outcome was the discovery of a diabetes after the OGTT test (75g of glucose), 2 to 3 months after delivery, a fasting blood glucose rate ≥ 1,26 g/L and a plasma glucose after 2 hours ≥ 2g/L

* In ERD2 study 391 subjects were included. The patients were over 18 years old and had a gestational diabetes and were informed by a survey. The main criteria of maternal and neonatal complications were a maternal high blood pressure, a neonatal jaundice, neonatal hypocalcemia and hypoglycemia, and shoulders dystocia. In this study the patients were followed up with classic diary for glycemic blood rate.
* With TELESUR-GDM study, the objective is to prove the non-inferiority of the new method of monitoring for blood glucose rate (myDiabby Healthcare) for patients who had a gestational diabetes and who gave birth between 01/01/2021 and the 31/12/2021. The data will be collected with an informatic secured data base.

ELIGIBILITY:
Inclusion Criteria :

* Age ≥18 years old
* Date of delivery between 01/01/2013 and 30/06/2015 Or
* Date of delivery between 01/01/2021 and 31/12/2021 and monitored by myDiabby Healthcare
* Patients who had a gestational diabetes tested according to CNGOF recommendations

Exclusion Criteria :

* Patients with type 2 or type 1 diabetes
* Opposition of the patient for participating to the study
* Patients who have had a multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women (≥ 18 years old) with gestational diabetes who gave birth between 01/01/2013 and 30/06/2015 for the control group (paper blood glucose diaries) or between 01/01/2021 and 31/12/2021 if they have benefited from remote monitoring with myDiabby Healthcare
Sampling Method: Non-Probability Sample
Enrollment: 668 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Assessment of the non-inferiority of the occurrence of maternal, fetal, and neonatal complications for patients of both groups | At the end of the Study, an average of 8 month
  Comparison, for patients with GDM, of the composite score (maternal / foetal - neonatal) between the group with remote monitoring by the myDiabby Healthcare and the group of patients with traditional monitoring (paper glycemic diaries). For each item answered "yes" count 1 point and "no" count 0 point.
  For information, the composite score is based on the following items:
  Maternal :
  * High blood pressure (≥140/90 mmHG)
  * Caesarean section
  * Instrumental extraction
  * Perineal Trauma : complete or complicated perineal tearing
  * Pre-eclampsia
  Foetal and neonatal :
  * birth weight ≥ 95th percentile for gestational age (neonatal macrosomia)
  * intrauterine growth restriction (birth weight ≤ 5th percentile)
  * APGAR < 7 at 5 minutes
  * Fetal death in utero
  * Neonatal hypoglycemia
  * Neonatal hypocalcemia
  * Neonatal acidosis : pH<7,10 and lactate >6µmol
  * Shoulders dystocia
  * Collarbone fracture, brachial plexus
  * Neonatal jaundice

SECONDARY OUTCOMES:
Comparison, for each maternal and each Foetal/Neonatal composite items, between both groups | At the end of the Study, an average of 8 month
  Prevalence of each maternal and each Foetal/Neonatal composite item in each group. For each item answered "yes" count 1 point and "no" count 0 point
  For information, the maternal composite items are as follows:
  * High blood pressure (≥140/90 mmHG)
  * Hospitalization during pregnancy
  * Caesarean section
  * Instrumental extraction
  * Perineal Trauma : complete or complicated perineal tearing
  * Pre-eclampsia
  For information, the Foetal/Neonatal composite items are as follows:
  * birth weight ≥ 95th percentile for gestational age (neonatal macrosomia)
  * intrauterine growth restriction (birth weight ≤ 5th percentile)
  * APGAR <7 at 5 minutes
  * Fetal death in utero
  * Neonatal hypoglycemia
  * Neonatal hypocalcemia
  * Neonatal acidosis : pH<7,10 and lactate >6µmol
  * Shoulders dystocia
  * Collarbone fracture, brachial plexus
  * Neonatal jaundice
Comparison of the rate of patients put on insulin in both groups | At the end of the Study, an average of 8 month
  Number of patients put on insulin in each group and comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Pr Christophe Poncelet, Principal Investigator — Hôpital NOVO; Dr Catherine Campinos, Principal Investigator — Hôpital NOVO
Locations (1):
- Endocrinology department - Centre Hospitalier René Dubos, Pontoise, France

IPD SHARING:
Plan to Share IPD: No